CLINICAL TRIAL: NCT04368728
Title: A PHASE 1/2/3, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND, DOSE-FINDING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, IMMUNOGENICITY, AND EFFICACY OF SARS-COV-2 RNA VACCINE CANDIDATES AGAINST COVID-19 IN HEALTHY INDIVIDUALS
Brief Title: Study to Describe the Safety, Tolerability, Immunogenicity, and Efficacy of RNA Vaccine Candidates Against COVID-19 in Healthy Individuals
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4591001; 2020-002641-42 (EudraCT Number)
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19; Coronavirus; Vaccine; SARS-CoV-2; RNA Vaccine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (20):
- 10 µg dose, 18-55 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 20 µg dose, 18-55 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 30 µg dose, 18-55 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 10 µg dose, 65-85 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 20 µg dose, 65-85 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 30 µg dose, 65-85 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1; Biological: BNT162b2
- 30 µg dose, ≥12 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b2
- Placebo, 18-55 years of age (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo, 65-85 years of age (Placebo Comparator)
  Interventions: Other: Placebo
- Placebo, ≥12 years of age (Placebo Comparator)
  Interventions: Other: Placebo
- 100 µg dose, 18-55 years of age (2 doses) (Experimental)
  Interventions: Biological: BNT162b1
- Vaccination of Placebo recipients with BNT162b2 - Stage 1 (Other): Participants ≥16 years of age who originally received placebo and are eligible for COVID-19 vaccination following any local or national recommendations will be offered the opportunity to receive BNT162b2 as part of the study.
  Interventions: Biological: BNT162b2
- Vaccination of placebo recipients with BNT162b2 - Stage 2 (Other): Participants ≥16 years of age who originally received placebo will be offered the opportunity to receive BNT162b2 at defined points as part of the study.
  Interventions: Biological: BNT162b2
- Booster vaccination of Phase 1 participants with BNT162b2 at a dose of 30 µg (Experimental)
  Interventions: Biological: BNT162b2
- Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 30 µg (Experimental)
  Interventions: Biological: BNT162b2
- Booster vaccination of Phase 3 participants with BNT162b2SA at a dose of 30 µg (Experimental)
  Interventions: Biological: BNT162b2SA
- Vaccination of BNT162b2-naive participants with BNT162b2SA at a dose of 30 µg (Experimental)
  Interventions: Biological: BNT162b2SA
- Booster and further vaccination of Phase 3 participants with BNT162b2SA at a dose of 30 µg (Experimental)
  Interventions: Biological: BNT162b2SA
- Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 5 µg (Experimental)
  Interventions: Biological: BNT162b2
- Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 10 µg (Experimental)
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b1 — Intramuscular injection
  Arms: 10 µg dose, 18-55 years of age (2 doses); 10 µg dose, 65-85 years of age (2 doses); 100 µg dose, 18-55 years of age (2 doses); 20 µg dose, 18-55 years of age (2 doses); 20 µg dose, 65-85 years of age (2 doses); 30 µg dose, 18-55 years of age (2 doses); 30 µg dose, 65-85 years of age (2 doses)
Biological: BNT162b2 — Intramuscular injection
  Arms: 10 µg dose, 18-55 years of age (2 doses); 10 µg dose, 65-85 years of age (2 doses); 20 µg dose, 18-55 years of age (2 doses); 20 µg dose, 65-85 years of age (2 doses); 30 µg dose, 18-55 years of age (2 doses); 30 µg dose, 65-85 years of age (2 doses); 30 µg dose, ≥12 years of age (2 doses); Booster vaccination of Phase 1 participants with BNT162b2 at a dose of 30 µg; Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 10 µg; Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 30 µg; Booster vaccination of Phase 3 participants with BNT162b2 at a dose of 5 µg; Vaccination of Placebo recipients with BNT162b2 - Stage 1; Vaccination of placebo recipients with BNT162b2 - Stage 2
Other: Placebo — Intramuscular injection
  Arms: Placebo, 18-55 years of age; Placebo, 65-85 years of age; Placebo, ≥12 years of age
Biological: BNT162b2SA — Intramuscular injection
  Arms: Booster and further vaccination of Phase 3 participants with BNT162b2SA at a dose of 30 µg; Booster vaccination of Phase 3 participants with BNT162b2SA at a dose of 30 µg; Vaccination of BNT162b2-naive participants with BNT162b2SA at a dose of 30 µg

SUMMARY:
This is a Phase 1/2/3, randomized, placebo-controlled, observer-blind, dose-finding, vaccine candidate-selection, and efficacy study in healthy individuals.

The study consists of 2 parts: Phase 1: to identify preferred vaccine candidate(s) and dose level(s); Phase 2/3: an expanded cohort and efficacy part.

The study will evaluate the safety, tolerability, and immunogenicity of 3 different SARS-CoV-2 RNA vaccine candidates against COVID-19 and the efficacy of 1 candidate:

* As a 2-dose (separated by 21 days) schedule;
* At various different dose levels in Phase 1;
* As a booster;
* In 3 age groups (Phase 1: 18 to 55 years of age, 65 to 85 years of age; Phase 2/3: ≥12 years of age [stratified as 12-15, 16-55 or >55 years of age]).

The candidate selected for efficacy evaluation in Phase 2/3 is BNT162b2 at a dose of 30 µg.

Participants who originally received placebo will be offered the opportunity to receive BNT162b2 at defined points as part of the study.

In order to describe the boostability of BNT162, and potential heterologous protection against emerging SARS-CoV-2 VOCs, an additional dose of BNT162b2 at 30 µg will be given to Phase 1 participants approximately 6 to 12 months after their second dose of BNT162b1 or BNT162b2. This will provide an early assessment of the safety of a third dose of BNT162, as well as its immunogenicity.

The assessment of boostability will be further expanded in a subset of Phase 3 participants at selected sites in the US who will receive a third dose of BNT162b2 at 30 µg or a third and potentially a fourth dose of prototype BNT162b2VOC at 30 µg (BNT162b2s01, based upon the South African variant and hereafter referred to as BNT162b2SA). A further subset of Phase 3 participants will receive a third, lower, dose of BNT162b2 at 5 or 10 µg.

To further describe potential homologous and heterologous protection against emerging SARS-CoV-2 VOCs, a new cohort of participants will be enrolled who are COVID-19 vaccine-naïve (ie, BNT162b2-naïve) and have not experienced COVID-19. They will receive BNT162b2SA given as a 2-dose series, separated by 21 days.

To reflect current and anticipated recommendations for COVID 19 vaccine boosters, participants in C4591001 who meet specified recommendations and have not already received one, will be offered a third dose of BNT162b2 after their second dose of BNT162.

ELIGIBILITY:
Inclusion Criteria:

• Male or female participants between the ages of 18 and 55 years, inclusive, 65 and 85 years, inclusive, or ≥12 years, inclusive, at randomization (dependent upon study phase). For the boostability and protection-against-VOCs subset: Existing participants enrolled to receive a third dose of BNT162b2 at 30 µg or BNT162b2SA; male or female participants between the ages of 18 and 55 years, inclusive, at rerandomization.

Newly enrolled participants enrolled to receive 2 doses of BNT162b2SA; male or female participants between the ages of 18 and 55 years, inclusive, at enrollment.

Existing participants enrolled to receive a third dose of BNT162b2 at 5 or 10 µg; male or female participants ≥18 years at rerandomization.

Note that participants <18 years of age cannot be enrolled in the EU.

* Participants who are willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
* Participants who, in the judgment of the investigator, are at risk for acquiring COVID-19.
* Boostability and protection-against-VOCs existing participant subset only: Participants who provided a serum sample at Visit 3, with Visit 3 occurring within the protocol-specified window.
* Capable of giving personal signed informed consent

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Phases 1 and 2 only: Known infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Receipt of medications intended to prevent COVID 19.
* Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID 19
* Phase 1 only: Individuals at high risk for severe COVID-19, including those with any of the following risk factors:

  * Hypertension
  * Diabetes mellitus
  * Chronic pulmonary disease
  * Asthma
  * Current vaping or smoking
  * History of chronic smoking within the prior year
  * BMI >30 kg/m2
  * Anticipating the need for immunosuppressive treatment within the next 6 months
* Phase 1 only: Individuals currently working in occupations with high risk of exposure to SARS-CoV-2 (eg, healthcare worker, emergency response personnel).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Phase 1 only: Individuals with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
* Women who are pregnant or breastfeeding.
* Previous vaccination with any coronavirus vaccine.
* Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study.
* Phase 1 only: Regular receipt of inhaled/nebulized corticosteroids.
* Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration or planned receipt throughout the study.
* Participation in other studies involving study intervention within 28 days prior to study entry through and including 6 months after the last dose of study intervention, with the exception of non-Pfizer interventional studies for prevention of COVID 19, which are prohibited throughout study participation.
* Previous participation in other studies involving study intervention containing lipid nanoparticles.
* Phase 1 only: Positive serological test for SARS-CoV-2 IgM and/or IgG antibodies at the screening visit.
* Phase 1 only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a ≥ Grade 1 abnormality.
* Phase 1 only: Positive test for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBc Abs), or hepatitis C virus antibodies (HCV Abs) at the screening visit.
* Phase 1 only: SARS-CoV-2 NAAT-positive nasal swab within 24 hours before receipt of study intervention.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47079 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants in Phase 1 reporting local reactions | For 7 days after dose 1 and dose 2
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
Percentage of participants in Phase 1 reporting systemic events | For 7 days after dose 1 and dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
Percentage of participants in Phase 1 reporting adverse events | From dose 1 through 1 month after the last dose
  As elicited by investigational site staff
Percentage of participants in Phase 1 reporting serious adverse events | From dose 1 through 6 months after the last dose
  As elicited by investigational site staff
Percentage of Phase 1 participants with abnormal hematology and chemistry laboratory values | 1 day after dose 1
  As measured at the central laboratory
Percentage of Phase 1 participants with abnormal hematology and chemistry laboratory values | 7 days after dose 1
  As measured at the central laboratory
Percentage of Phase 1 participants with abnormal hematology and chemistry laboratory values | 7 days after dose 2
  As measured at the central laboratory
Percentage of Phase 1 participants with grading shifts in hematology and chemistry laboratory assessments | Between baseline and 1 day after dose 1
  As measured at the central laboratory
Percentage of Phase 1 participants with grading shifts in hematology and chemistry laboratory assessments | Between baseline and 7 days after dose 1
  As measured at the central laboratory
Percentage of Phase 1 participants with grading shifts in hematology and chemistry laboratory assessments | Between before dose 2 and 7 days after dose 2
  As measured at the central laboratory
In the first 360 participants randomized into Phase 2/3, percentage of participants reporting local reactions | For 7 days after dose 1 and dose 2
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
In the first 360 participants randomized into Phase 2/3, percentage of participants reporting systemic events | For 7 days after dose 1 and dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
In the first 360 participants randomized into Phase 2/3, percentage of participants reporting adverse events | From dose 1 through 1 month after the last dose
  As elicited by investigational site staff
In the first 360 participants randomized into Phase 2/3, percentage of participants reporting serious adverse events | From dose 1 through 6 months after the last dose
  As elicited by investigational site staff
In a subset of at least 6000 participants randomized in Phase 2/3, percentage of participants reporting local reactions | For 7 days after dose 1 and dose 2
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
In a subset of at least 6000 participants randomized in Phase 2/3, percentage of participants reporting systemic events | For 7 days after dose 1 and dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
Percentage of participants in Phase 2/3 reporting adverse events | From dose 1 through 1 month after the last dose
  As elicited by investigational site staff
Percentage of participants in Phase 2/3 reporting serious adverse events | From dose 1 through 6 months after the last dose
  As elicited by investigational site staff
Confirmed COVID-19 in Phase 2/3 participants without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 in Phase 2/3 participants with and without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Percentage of participants 12-15 years of age in Phase 3 reporting adverse events | From dose 1 through 1 month after the last dose
  As elicited by investigational site staff
Percentage of participants 12-15 years of age in Phase 3 reporting adverse events | From dose 1 through 6 months after the last dose
  As elicited by investigational site staff
In participants 12-15 years of age randomized in Phase 3, percentage of participants reporting local reactions | For 7 days after dose 1 and dose 2
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
In participants 12-15 years of age randomized in Phase 3, percentage of participants reporting systemic events | For 7 days after dose 1 and dose 2
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
In participants who receive BNT162b2SA given as 1 or 2 doses, percentage of participants reporting adverse events | From dose 1 through 1 month after the last dose
  As elicited by investigational site staff
In participants who receive BNT162b2SA given as 1 or 2 doses, percentage of participants reporting serious adverse events | From dose 1 through 5 or 6 months after the last dose
  As elicited by investigational site staff
In participants, who receive BNT162b2SA given as 1 or 2 doses, percentage of participants reporting local reactions | For 7 days after dose 1 (and dose 2)
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
In participants who receive BNT162b2SA given as 1 or 2 doses, percentage of participants reporting systemic events | For 7 days after dose 1 (and dose 2)
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
In participants who receive a third dose of BNT162b2 as part of the subset for evaluation of boostability and protection against emerging VOCs, percentage of participants reporting adverse events | From the third dose through 1 month after the third dose
  As elicited by investigational site staff
In participants who receive a third dose of BNT162b2 as part of the subset for evaluation of boostability and protection against emerging VOCs, percentage of participants reporting serious adverse events | From the third dose through 6 months after the third dose
  As elicited by investigational site staff
In participants who receive a third dose of BNT162b2 as part of the subset for evaluation of boostability and protection against emerging VOCs, percentage of participants reporting local reactions | For 7 days after the third dose
  Pain at the injection site, redness, and swelling as self-reported on electronic diaries.
In participants who receive a third dose of BNT162b2 as part of the subset for evaluation of boostability and protection against emerging VOCs, percentage of participants reporting systemic events | For 7 days after the third dose
  Fever, fatigue, headache, chills, vomiting, diarrhea, new or worsened muscle pain, and new or worsened joint pain as self-reported on electronic diaries.
In participants who receive a third dose of BNT162b2 as a result of current or anticipated recommendations, percentage of participants reporting adverse events | From the third dose through 1 month after the third dose
  As elicited by investigational site staff
In participants who receive a third dose of BNT162b2 as a result of current or anticipated recommendations, percentage of participants reporting serious adverse events | From the third dose through 6 months after the third dose
  As elicited by investigational site staff
Noninferiority of the SARS-CoV-2 reference strain neutralizing titers after a third dose of BNT162b2 at 30 µg compared to after 2 doses of BNT162b2, in the same individuals | 1 month after the third dose
  As measured at the central laboratory
Noninferiority of the SARS-CoV-2 SA strain neutralizing titers after one dose of BNT162b2SA compared to the SARS-CoV-2 reference strain neutralizing titers after 2 doses of BNT162b2, in the same individuals | 1 month after the third dose
  As measured at the central laboratory
Noninferiority of the SARS-CoV-2 SA strain neutralizing titers after 2 doses of BNT162b2SA compared to the SARS-CoV-2 reference strain neutralizing titers after 2 doses of BNT162b2 | 1 month after the second dose
  As measured at the central laboratory

SECONDARY OUTCOMES:
In Phase 1 participants, SARS-CoV-2 serum neutralizing antibody levels, expressed as GMTs | Through 2 years after the final dose
  As measured at the central laboratory
In Phase 1 participants, GMFR in SARS-CoV-2 serum neutralizing titers from before vaccination to each subsequent time point | Through 2 years after the final dose
  As measured at the central laboratory
Proportion of participants in Phase 1 achieving a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2 serum neutralizing antibody levels | Through 2 years after the final dose
  As measured at the central laboratory
In Phase 1 participants, SARS-CoV-2 anti-S1 binding antibody levels and anti-RBD binding antibody levels, expressed as GMCs | Through 2 years after the final dose
  As measured at the central laboratory
Proportion of participants in Phase 1 achieving a greater than or equal to 4-fold rise from before vaccination in SARS-CoV-2 anti-S1 binding antibody levels and anti-RBD binding antibody levels | Through 2 years after the final dose
  As measured at the central laboratory
In Phase 1 participants, GMFR in SARS-CoV-2 anti-S1 binding antibody levels and anti-RBD binding antibody levels from before vaccination to each subsequent time point | Through 2 years after the final dose
  As measured at the central laboratory
In Phase 1 participants, GMR of the geometric mean of SARS-CoV-2 serum neutralizing titers to the geometric mean of SARS CoV 2 (anti-S1 and anti-RBD) binding antibody levels | Through 2 years after the final dose
  As measured at the central laboratory
Confirmed COVID-19 in Phase 2/3 participants without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 in Phase 2/3 participants with and without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed severe COVID-19 in Phase 2/3 participants without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed severe COVID-19 in Phase 2/3 participants without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed severe COVID-19 in Phase 2/3 participants with and without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed severe COVID-19 in Phase 2/3 participants with and without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 (according to the CDC-defined symptoms) in Phase 2/3 participants without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 (according to the CDC-defined symptoms) in Phase 2/3 participants without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 (according to the CDC-defined symptoms) in Phase 2/3 participants with and without evidence of infection before vaccination | From 7 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
Confirmed COVID-19 (according to the CDC-defined symptoms) in Phase 2/3 participants with and without evidence of infection before vaccination | From 14 days after the second dose of study intervention to the end of the study, up to 2 years
  Per 1000 person-years of follow-up
GMR of SARS CoV 2 neutralizing titers in the 2 age groups (12-15 years of age to 16-25 years of age) | 1 month after the second dose
  As measured at the central laboratory
Incidence of asymptomatic SARS CoV-2 infection based on N binding antibody seroconversion in participants with no serological or virological evidence of past SARS CoV-2 infection or confirmed COVID-19 prior to 1 month after receipt of the second dose | Through 1 month after the second dose
  Per 1000 person-years of follow-up
Incidence of asymptomatic SARS CoV-2 infection based on central laboratory-confirmed NAAT in participants with no serological or virological evidence (up to the start of the asymptomatic surveillance period) of past SARS-CoV-2 infection | Through 6 months after the second dose
  Per 1000 person-years of follow-up
Noninferiority of the SARS-CoV-2 SA strain neutralizing titers after a third dose of BNT162b2 at 30 µg compared to the SARS-CoV-2 reference strain neutralizing titers after 2 doses of BNT162b2, in the same individuals | 1 month after the third dose
  As measured at the central laboratory
Noninferiority of the SARS-CoV-2 reference strain neutralizing titers after one dose of BNT162b2SA compared to after 2 doses of BNT162b2, in the same individuals | 1 month after the first dose of BNT162b2SA
  As measured at the central laboratory
Comparison of the SARS-CoV-2 SA strain neutralizing titers after 1 dose of BNT162b2SA to after a third dose of BNT162b2 at 30 µg | 1 month after the first dose of BNT162b2SA/third dose of BNT162b2
  As measured at the central laboratory
Comparison of the SARS-CoV-2 SA strain neutralizing titers after 2 doses of BNT162b2SA to the SARS-CoV-2 reference strain neutralizing titers after 2 doses of BNT162b2, in the same individuals | 1 month after the second dose of BNT162b2SA
  As measured at the central laboratory
Comparison of the SARS-CoV-2 SA strain neutralizing titers after 2 doses of BNT162b2SA to after 2 doses of BNT162b2 | 1 month after the second dose
  As measured at the central laboratory
Comparison of the SARS-CoV-2 reference strain neutralizing titers after 2 doses of BNT162b2SA to after 2 doses of BNT162b2 | 1 month after the second dose
  As measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (167):
- United States (145):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Birmingham Clinical Research Unit, Birmingham, Alabama
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Optimal Research, LLC, Huntsville, Alabama
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - Chinle Comprehensive Health Care Facility, Chinle, Arizona
  - Johns Hopkins Center for American Indian Health, Chinle, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Whiteriver Indian Hospital, Whiteriver, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Long Beach Clinical Trials Services Inc., Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Paradigm Clinical Research Center, Redding, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - Clinical and Translational Science Center (CTSC) Clinical Research Center (CCRC), Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - California Research Foundation, San Diego, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Bayview Research Group, Valley Village, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Lynn Institute of Denver, Aurora, Colorado
  - Clinical Research Consulting, LLC, Milford, Connecticut
  - Yale Center for Clinical Investigations (CSRU), New Haven, Connecticut
  - Alliance for Multispecialty Research, Coral Gables, Florida
  - DeLand Clinical Research Unit, DeLand, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - IACT Health, Columbus, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Solaris Clinical Research, Meridian, Idaho
  - Optimal Research, Peoria, Illinois
  - University of Iowa Hospitals & Clinics Investigational Drug Servces, Iowa City, Iowa
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport Clinical Trials Office, Shreveport, Louisiana
  - LSUHSC-Shreveport, Shreveport, Louisiana
  - Pharmaron CPC, Inc., Baltimore, Maryland
  - University of Maryland Medical Center Investigational Drug Service Pharmacy, Baltimore, Maryland
  - University of Maryland, Baltimore, Health Sciences Research Facility III, Baltimore, Maryland
  - University of Maryland, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Michigan Center for Medical Research, Farmington Hills, Michigan
  - MedPharmics, LLC, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Bozeman Health Deaconess Hospital dba Bozeman Health Clinical Research, Bozeman, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Methodist Physicians Clinic / CCT Research, Fremont, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Wake Research-Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Amici Clinical Research, Raritan, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Johns Hopkins Center for American Indian Health, Gallup, New Mexico
  - Johns Hopkins Center for American Indian Health, Shiprock, New Mexico
  - Meridian Clinical Research, LLC, Binghamton, New York
  - Meridian Clinical Research LLC, Endwell, New York
  - NYU Langone Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - University of Rochester Medical Center- Kari Steinmetz, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Global Health Research Unit, Syracuse, New York
  - Meridian Clinical Research LLC, Vestal, New York
  - PMG Research of Raleigh, LLC d/b/a PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte LLC, Charlotte, North Carolina
  - Accessioning Unit and Repository, Durham, North Carolina
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Clinical Research Pickett Road, Durham, North Carolina
  - Duke Investigational Drug Service Pharmacy, Durham, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Lillestol Research Llc, Fargo, North Dakota
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Meridian Clinical Research LLC, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - VA Northeast Ohio Healthcare System, Cleveland, Ohio
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Kaiser Permanente Northwest-Center for Health Research, Portland, Oregon
  - Lehigh Valley Health Network/Network Office of Research and Innovation, Allentown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Main Street Physician's Care, Little River, South Carolina
  - Main Street Physician's Care, Loris, South Carolina
  - Holston Medical Group, Bristol, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Trinity Clinical Research, Tullahoma, Tennessee
  - Benchmark Research, Austin, Texas
  - ARC Clinical Research at Four Points, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Tekton Research, Austin, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Resources, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Ventavia Research Group, LLC, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Ventavia Research Group, LLC, Keller, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Benchmark Research., San Angelo, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Virginia Research Center LLC, Midlothian, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Wenatchee Valley Hospital, Wenatchee, Washington
- Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, CABA, Argentina
- Brazil (2):
  - Hospital Santo Antonio/ Associacao Obras Sociais Irma Dulce, Salvador, Estado de Bahia
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda (Casa Branca), São Paulo
- Germany (6):
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - Medizentrum Essen Borbeck, Essen
  - IKF Pneumologie GmbH & Co KG, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - CRS Clinical Research Services Mannheim GmbH, Mannheim
  - Studienzentrum Brinkum Dr. Lars Pohlmeier und Torsten Drescher, Stuhr
- South Africa (4):
  - Newtown Clinical Research Centre, Johannesburg, Gauteng
  - Jongaie Research, Pretoria, Gauteng
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Tiervlei Trial Centre, Basement Level, Karl Bremer Hospital, Cape Town, Western Cape
- Turkey (Türkiye) (9):
  - Ankara Universitesi Tip Fakultesi, Ibni Sina Hastanesi, Ankara
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Istanbul Yedikule Gogus Hastaliklari ve Gogus Cerrahisi Egitim Arastirma Hastanesi, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi-Cerrahpasa, Cerrahpasa Tip Fakultesi, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - Acibadem Atakent Hastanesi, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi, Sakarya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463
- [Derived] Pather S, Charpentier N, van den Ouweland F, Rizzi R, Finlayson A, Salisch N, Muik A, Lindemann C, Khanim R, Abduljawad S, Smith ER, Gurwith M, Chen RT; Benefit-Risk Assessment of VAccines by TechnolOgy Working Group (BRAVATO; ex-V3SWG). A Brighton Collaboration standardized template with key considerations for a benefit-risk assessment for the Comirnaty COVID-19 mRNA vaccine. Vaccine. 2024 Sep 17;42(22):126165. doi: 10.1016/j.vaccine.2024.126165. Epub 2024 Aug 27. PMID 39197299
- [Derived] Killeen T, Kermer V, Troxler Saxer R. mRNA vaccine development during the COVID-19 pandemic: a retrospective review from the perspective of the Swiss affiliate of a global biopharmaceutical company. J Pharm Policy Pract. 2023 Nov 27;16(1):158. doi: 10.1186/s40545-023-00652-y. PMID 38012751
- [Derived] Fraiman J, Erviti J, Jones M, Greenland S, Whelan P, Kaplan RM, Doshi P. Serious adverse events of special interest following mRNA COVID-19 vaccination in randomized trials in adults. Vaccine. 2022 Sep 22;40(40):5798-5805. doi: 10.1016/j.vaccine.2022.08.036. Epub 2022 Aug 31. PMID 36055877
- [Derived] Kurhade C, Zou J, Xia H, Liu M, Yang Q, Cutler M, Cooper D, Muik A, Sahin U, Jansen KU, Ren P, Xie X, Swanson KA, Shi PY. Neutralization of Omicron sublineages and Deltacron SARS-CoV-2 by three doses of BNT162b2 vaccine or BA.1 infection. Emerg Microbes Infect. 2022 Dec;11(1):1828-1832. doi: 10.1080/22221751.2022.2099305. PMID 35792746
- [Derived] Kurhade C, Zou J, Xia H, Cai H, Yang Q, Cutler M, Cooper D, Muik A, Jansen KU, Xie X, Swanson KA, Shi PY. Neutralization of Omicron BA.1, BA.2, and BA.3 SARS-CoV-2 by 3 doses of BNT162b2 vaccine. Nat Commun. 2022 Jun 23;13(1):3602. doi: 10.1038/s41467-022-30681-1. PMID 35739094
- [Derived] De Santis F, Gubbiotti S. Borrowing historical information for non-inferiority trials on Covid-19 vaccines. Int J Biostat. 2022 Apr 27;19(1):177-189. doi: 10.1515/ijb-2021-0120. eCollection 2023 May 1. PMID 35472295
- [Derived] Thomas SJ, Perez JL, Lockhart SP, Hariharan S, Kitchin N, Bailey R, Liau K, Lagkadinou E, Tureci O, Sahin U, Xu X, Koury K, Dychter SS, Lu C, Gentile TC, Gruber WC. Efficacy and safety of the BNT162b2 mRNA COVID-19 vaccine in participants with a history of cancer: subgroup analysis of a global phase 3 randomized clinical trial. Vaccine. 2022 Mar 1;40(10):1483-1492. doi: 10.1016/j.vaccine.2021.12.046. Epub 2021 Dec 24. PMID 35131133
- [Derived] Thomas SJ, Moreira ED Jr, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Polack FP, Zerbini C, Bailey R, Swanson KA, Xu X, Roychoudhury S, Koury K, Bouguermouh S, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Yang Q, Liberator P, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Gruber WC, Jansen KU; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine through 6 Months. N Engl J Med. 2021 Nov 4;385(19):1761-1773. doi: 10.1056/NEJMoa2110345. Epub 2021 Sep 15. PMID 34525277
- [Derived] Frenck RW Jr, Klein NP, Kitchin N, Gurtman A, Absalon J, Lockhart S, Perez JL, Walter EB, Senders S, Bailey R, Swanson KA, Ma H, Xu X, Koury K, Kalina WV, Cooper D, Jennings T, Brandon DM, Thomas SJ, Tureci O, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety, Immunogenicity, and Efficacy of the BNT162b2 Covid-19 Vaccine in Adolescents. N Engl J Med. 2021 Jul 15;385(3):239-250. doi: 10.1056/NEJMoa2107456. Epub 2021 May 27. PMID 34043894
- [Derived] Vogel AB, Kanevsky I, Che Y, Swanson KA, Muik A, Vormehr M, Kranz LM, Walzer KC, Hein S, Guler A, Loschko J, Maddur MS, Ota-Setlik A, Tompkins K, Cole J, Lui BG, Ziegenhals T, Plaschke A, Eisel D, Dany SC, Fesser S, Erbar S, Bates F, Schneider D, Jesionek B, Sanger B, Wallisch AK, Feuchter Y, Junginger H, Krumm SA, Heinen AP, Adams-Quack P, Schlereth J, Schille S, Kroner C, de la Caridad Guimil Garcia R, Hiller T, Fischer L, Sellers RS, Choudhary S, Gonzalez O, Vascotto F, Gutman MR, Fontenot JA, Hall-Ursone S, Brasky K, Griffor MC, Han S, Su AAH, Lees JA, Nedoma NL, Mashalidis EH, Sahasrabudhe PV, Tan CY, Pavliakova D, Singh G, Fontes-Garfias C, Pride M, Scully IL, Ciolino T, Obregon J, Gazi M, Carrion R Jr, Alfson KJ, Kalina WV, Kaushal D, Shi PY, Klamp T, Rosenbaum C, Kuhn AN, Tureci O, Dormitzer PR, Jansen KU, Sahin U. BNT162b vaccines protect rhesus macaques from SARS-CoV-2. Nature. 2021 Apr;592(7853):283-289. doi: 10.1038/s41586-021-03275-y. Epub 2021 Feb 1. PMID 33524990
- [Derived] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246
- [Derived] Walsh EE, Frenck RW Jr, Falsey AR, Kitchin N, Absalon J, Gurtman A, Lockhart S, Neuzil K, Mulligan MJ, Bailey R, Swanson KA, Li P, Koury K, Kalina W, Cooper D, Fontes-Garfias C, Shi PY, Tureci O, Tompkins KR, Lyke KE, Raabe V, Dormitzer PR, Jansen KU, Sahin U, Gruber WC. Safety and Immunogenicity of Two RNA-Based Covid-19 Vaccine Candidates. N Engl J Med. 2020 Dec 17;383(25):2439-2450. doi: 10.1056/NEJMoa2027906. Epub 2020 Oct 14. PMID 33053279
- [Derived] Mulligan MJ, Lyke KE, Kitchin N, Absalon J, Gurtman A, Lockhart S, Neuzil K, Raabe V, Bailey R, Swanson KA, Li P, Koury K, Kalina W, Cooper D, Fontes-Garfias C, Shi PY, Tureci O, Tompkins KR, Walsh EE, Frenck R, Falsey AR, Dormitzer PR, Gruber WC, Sahin U, Jansen KU. Phase I/II study of COVID-19 RNA vaccine BNT162b1 in adults. Nature. 2020 Oct;586(7830):589-593. doi: 10.1038/s41586-020-2639-4. Epub 2020 Aug 12. PMID 32785213
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591001